CLINICAL TRIAL: NCT06052124
Title: Merging Augmented Reality and Neuroimaging to Improve Patient Safety and Outcomes for Neurosurgical Procedures
Brief Title: Augmented Reality for Subdural Drain Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vivek P. Buch, Assistant Clinical Professor of Neurosurgery, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 70606
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Pilot Usability (Part 1) (Experimental): Five patients will be enrolled to test whether the AR device functions appropriately, but no clinical decisions or changes to care will be determine by the AR device at this point.
  Interventions: Device: Augmented Reality Device
- AR Guided SEPS Placement (Part 2) (Experimental): AR guidance is used to place SEPS drain
  Interventions: Device: Augmented Reality Device
- Anatomical Guided SEPS Placement (Part 2) (No Intervention): Standard of care, non AR guided SEPS drain placement

INTERVENTIONS:
Device: Augmented Reality Device — AR device will be used to determine where to place SEPS drain
  Arms: AR Guided SEPS Placement (Part 2); Pilot Usability (Part 1)

SUMMARY:
This study involves using a augmented reality (AR) system to assist in the placement of a subdural evacuating portal system (SEPS). In the first part of the study, all participants will have skin marking of an AR-guided and non-AR-guided site to determine feasibility and method accuracy. In the second part, subjects will be randomized to AR-guided and non-AR-guided SEPS placement to determine efficacy.

DETAILED DESCRIPTION:
Chronic/subacute subdural hematoma (SDH) is one of the most common diseases encountered in neurosurgical practice. However, there is little consensus on first-line treatment. The SEPS was developed to implement a minimally invasive approach to drainage. New imaging technologies, such as augmented reality (AR) interfaces, can provide anatomical models and can help visualize hidden structures. The hope is that this study can give insight on whether AR-guidance can be used to improve SEPS placement, which can lead to higher volume drainage, greater symptomatic improvement, and decreased hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or Bilateral subdural hematoma that is planned to be treated by SEPS

Exclusion Criteria

* Unable to have CT scan
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean accuracy (in mm) of SEPS placement | Intra-procedural and up to 24 hours post procedure
  Comparison of measurements obtained by standard of care surface measurements and placement using AR guidance, and post placement CT scans.

SECONDARY OUTCOMES:
Change in size (mm) of subdural hematoma | Pre-procedure and 24 hours after SEPS placement
  Radiographic measure of thickest hematoma volume in sagittal and coronal planes after subdural evacuation compared to pre-procedure imaging, assessed in the randomized AR-guided and non-AR-guided arms only.
Change in symptom score | Assess at 24 hours status post SEPS placement and again at 1 month
  Composite measure, scaled from 0 (no symptoms) to 10 (severe symptoms), scored by clinician based overall impression of objective and subjective signs and symptoms including neurological strength exam, cognitive status, and patient self-reported symptomatic change, assessed in the randomized AR-guided and non-AR-guided arms only.
Length of hospital stay | Approximately 2 to 5 days
  Number of days since procedure between SEPS placement and discharge from inpatient stay, assessed in the randomized AR-guided and non-AR-guided arms only.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek P Buch, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No